CLINICAL TRIAL: NCT06742853
Title: A Phase 1, Randomized, Single-blind, Placebo-controlled Study to Investigate the Pharmacokinetics, Safety, Tolerability, and Efficacy of AZD0780 in Combination With Ezetimibe, Ezetimibe/Rosuvastatin, or Ezetimibe/Bempedoic Acid in Healthy Male and Female Participants 18 to 75 Years of Age With Elevated LDL-C.
Brief Title: A Study to Investigate the Pharmacokinetics, Safety, Tolerability, and Efficacy of AZD0780 With Ezetimibe Combinations in Healthy Adults With Elevated LDL-C.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7960C00017
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Dyslipidemia
Keywords: LDL-C; Hypercholesterolemia; Cholesterol absorption inhibitor; ATP-citrate lyase inhibitor
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — Ezetimibe; Rosuvastatin Calcium; 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Ezetimibe + AZD0780 (Experimental): Participants will receive ezetimibe 10 mg and AZD0780 once daily (QD) for 4 weeks.
  Interventions: Drug: AZD0780; Drug: Ezetimibe
- Rosuvastatin + Ezetimibe + AZD0780 (Experimental): Participants will receive rosuvastatin 20 mg, ezetimibe 10 mg and AZD0780 QD for 4 weeks.
  Interventions: Drug: AZD0780; Drug: Ezetimibe; Drug: Rosuvastatin
- Bempedoic Acid + Ezetimibe + AZD0780 (Optional Cohort) (Experimental): Participants will receive bempedoic acid 180 mg, ezetimibe 10 mg and AZD0780 QD for 4 weeks.
  Interventions: Drug: AZD0780; Drug: Ezetimibe; Drug: Bempedoic Acid
- Ezetimibe + Placebo (Placebo Comparator): Participants will receive ezetimibe 10 mg and placebo QD for 4 weeks.
  Interventions: Drug: Ezetimibe; Drug: Placebo
- Rosuvastatin + Ezetimibe + Placebo (Placebo Comparator): Participants will receive rosuvastatin 20 mg, ezetimibe 10 mg and placebo QD for 4 weeks.
  Interventions: Drug: Ezetimibe; Drug: Rosuvastatin; Drug: Placebo
- Bempedoic Acid + Ezetimibe + Placebo (Optional Cohort) (Placebo Comparator): Participants will receive bempedoic acid 180 mg, ezetimibe 10 mg and placebo QD for 4 weeks.
  Interventions: Drug: Ezetimibe; Drug: Bempedoic Acid; Drug: Placebo

INTERVENTIONS:
Drug: AZD0780 — AZD0780 tablet will be administered orally.
  Arms: Bempedoic Acid + Ezetimibe + AZD0780 (Optional Cohort); Ezetimibe + AZD0780; Rosuvastatin + Ezetimibe + AZD0780
Drug: Ezetimibe — Ezetimibe tablet will be administered orally.
Drug: Rosuvastatin — Rosuvastatin tablet will be administered orally.
  Arms: Rosuvastatin + Ezetimibe + AZD0780; Rosuvastatin + Ezetimibe + Placebo
Drug: Bempedoic Acid — Bempedoic Acid tablet will be administered orally.
  Arms: Bempedoic Acid + Ezetimibe + AZD0780 (Optional Cohort); Bempedoic Acid + Ezetimibe + Placebo (Optional Cohort)
Drug: Placebo — Placebo will be administered orally.
  Arms: Bempedoic Acid + Ezetimibe + Placebo (Optional Cohort); Ezetimibe + Placebo; Rosuvastatin + Ezetimibe + Placebo

SUMMARY:
The main aim of this study is to assess the effects of AZD0780 when added on top of ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled study in healthy participants with elevated low-density lipoprotein-cholesterol (LDL-C).

This study will assess the pharmacokinetic (PK), safety, tolerability, and efficacy of AZD0780 in combination with ezetimibe, ezetimibe/rosuvastatin, and ezetimibe/bempedoic acid.

Participants will be randomized to receive either AZD0780 or placebo (to be administered with ezetimibe, ezetimibe/rosuvastatin, or ezetimibe/bempedoic acid).

The study will comprise:

1. A Screening Period of up to 28 days.
2. A Run-in Period of 28 days.
3. A Treatment Period of 28 days.
4. Two Follow-up Visits, one and two weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form before any study-related procedure.
2. All females must have a negative serum pregnancy test at the Screening Visit and on admission to the Clinical Unit
3. Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria: postmenopausal or surgically sterilized females.
4. Have a Body Mass Index (BMI) > 18 kg/m² and weigh at least 50 kg.
5. Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.
6. Fasting LDL-C > 100 mg/dL but < 190 mg/dL (> 2.6 mmol/L but < 4.9 mmol/L for London EPCU) at the Screening Visit.
7. Fasting triglycerides < 400 mg/dL (or < 10.3 mmol/L for London EPCU) at the Screening Visit.

Exclusion Criteria:

1. History of any clinically important disease or disorder.
2. History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
4. Any laboratory values with specific deviations in alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin (TBL), estimated glomerular filtration rate, or hemoglobin at the Screening Visit or on Admission
5. Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results other than those described under exclusion criterion number 4, at Screening and/or Admission to the Clinical Unit
6. Any positive result on Screening for serum HBsAg, hepatitis B core antibody or human immunodeficiency virus.
7. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0780, ezetimibe, rosuvastatin, and bempedoic acid.
8. Treatment with any lipid-lowering therapy or AZD0780 within the 3 months prior to Screening.
9. Treatment with drugs for reduction or inhibition of Proprotein convertase subtilisin/kexin type 9 (PCSK9) within the last 12 months prior to Screening (approved or investigational and apart from AZD0780).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in direct Low-density Lipsprotein Cholesterol (LDL-C) | Week 4
  To evaluate the effect of AZD0780 on LDL-C levels versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Number of participants with adverse events | From screening (Day -56 to -29) to 14 Weeks
  The safety and tolerability of AZD0780 when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid will be assessed.

SECONDARY OUTCOMES:
Plasma concentration of AZD0780 | From Day 1 to Day 42
  To further characterize AZD0780 pharmacokinetics (PK) in plasma.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | From Day 1 to Day 42
  To further characterize AZD0780 PK in plasma.
Area under concentration-time curve in the dosing interval (AUCtau) (Day 15) | From Day 1 to Day 42
  To further characterize AZD0780 PK in plasma.
Maximum observed drug concentration (Cmax) | From Day 1 to Day 42
  To further characterize AZD0780 PK in plasma.
Time to reach maximum observed concentration (tmax) | From Day 1 to Day 42
  To further characterize AZD0780 PK in plasma.
Change from baseline in LDL-C ultra | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in LDL-C Friedewald | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in total cholesterol | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in non- HDL-C (high-density lipoprotein-cholesterol) | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in HDL-C | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in triglycerides | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in in Lipoprotein A [Lp(a)] | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.
Change from baseline in Apolipoprotein B (ApoB) | Week 4
  To evaluate the effect of AZD0780 on lipid parameters and inflammatory markers versus placebo when dosed with ezetimibe or ezetimibe and rosuvastatin or ezetimibe and bempedoic acid.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/